CLINICAL TRIAL: NCT03522532
Title: Redox Interactions Between Dental Restorations and Gingival Crevicular Fluid
Brief Title: Dental Restorations Effect on Oxidative Status of the Gingival Crevicular Fluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ervin Taso (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Sponsor-Investigator, Ervin Taso, Principal Investigator, Military Medical Academy, Belgrade, Serbia
Organization: Military Medical Academy, Belgrade, Serbia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VMA/10-12/A.1
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Pharmacological Action
Keywords: dental restorations; gingival crevicular fluid; glutathione; lipid peroxidation; superoxide dismutase

STUDY DESIGN:
Intervention Model Description: According to Black's Classification Criteria, patients were classified into four groups (K2 - K5). The number of patients within those groups were as follows: K2 (n=58), K3 (n=10), K4 (n=6) and K5 (n=14).
  Six different DMs were used in this study. The type of DM to be used for each patient was determined in relation to the dental lesion degree. DM placement was performed in one session and only one type was used per patient. Accordingly, 6 groups (arms) of dental patients (Amg, ZnPhC, ZnPoC, GIC, TEC and BF) were formed.
  Parameters of OS (MDA, GSH and tSOD) were measured in the GCF of the patients both before (day 0) and after treatment (on the 7th and 30th day).
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Amalgam (Amg) (Experimental): Amalgam was sealed in 8-K2 patients and 6-K2 patients. Oxidative stress parameters (MDA, GSH, tSOD) were measured in GCF prior to treatment and on the 7th and 30th day after treatment.
  Interventions: Procedure: Amalgam placement
- Tetric EvoCeram (TEC) (Experimental): Tetric EvoCeram was sealed in 12-K2 patients and 5-K5 patients. Oxidative stress parameters (MDA, GSH, tSOD) were measured in GCF prior to treatment and on the 7th and 30th day after treatment.
  Interventions: Procedure: Tetric EvoCeram placement
- Beautifil (BF) (Experimental): Beautifil was sealed in 15-K2 patients. Oxidative stress parameters (MDA, GSH, tSOD) were measured in GCF prior to treatment and on the 7th and 30th day after treatment.
  Interventions: Procedure: Beautifil placement
- Zinc phosphate cement (ZPhC) (Experimental): Zinc phosphate cement was sealed in 7-K2 patients, 4-K3 patients, 1-K4 patients and 2-K5 patients.
  Oxidative stress parameters (MDA, GSH, tSOD) were measured in GCF prior to treatment and on the 7th and 30th day after treatment.
  Interventions: Procedure: Zinc phosphate cement placement
- Zinc polycarboxylate cement (ZPoC) (Experimental): Zinc polycarboxylate cement was sealed in 5-K2 patients, 4-K3 patients and 5-K4 patients.
  Oxidative stress parameters (MDA, GSH, tSOD) were measured in GCF prior to treatment and on the 7th and 30th day after treatment.
  Interventions: Procedure: Zinc polycarboxylate cement placement
- Glass ionomer cement (GIC) (Experimental): Glass ionomer cement was sealed in 11-K2 patients, 2-K3 patients and 1-K5 patients.
  Oxidative stress parameters (MDA, GSH, tSOD) were measured in GCF prior to treatment and on the 7th and 30th day after treatment.
  Interventions: Procedure: Glass ionomer cement placement

INTERVENTIONS:
Procedure: Amalgam placement — Before the Amg was sealed GCF was taken, and then taken again on the 7th and 30th days after the applied treatment.
  Arms: Amalgam (Amg)
Procedure: Tetric EvoCeram placement — Before the TEC was sealed GCF was taken, and then taken again on the 7th and 30th days after the applied treatment.
  Arms: Tetric EvoCeram (TEC)
Procedure: Beautifil placement — Before the BF was sealed GCF was taken, and then taken again on the 7th and 30th days after the applied treatment.
  Arms: Beautifil (BF)
Procedure: Zinc phosphate cement placement — Before the ZPhC was sealed GCF was taken, and then taken again on the 7th and 30th days after the applied treatment.
  Arms: Zinc phosphate cement (ZPhC)
Procedure: Zinc polycarboxylate cement placement — Before the ZPoC was sealed GCF was taken, and then taken again on the 7th and 30th days after the applied treatment.
  Arms: Zinc polycarboxylate cement (ZPoC)
Procedure: Glass ionomer cement placement — Before the GIC was sealed GCF was taken, and then taken again on the 7th and 30th days after the applied treatment.
  Arms: Glass ionomer cement (GIC)

SUMMARY:
The goal of the study was to ascertain the influence of dental caries and teeth position as well as the type and amount of the applied dental materials (DMs) on the oxidative stress (OS) status in gingival crevicular fluid (GCF).

DETAILED DESCRIPTION:
Six DMs were tested by investigators, each sealed in one session: amalgam (Amg), zinc phosphate cement (ZnPhC), zinc polycarboxylate cement (ZnPoC), glass ionomer cement (GIC) and composites, Tetric EvoCeram (TEC) and Beautifil (BF).

The study included 88 dental outpatients. Oxidative stress parameters, including malondialdehyde (MDA), glutathione (GSH) and total superoxide dismutase (tSOD) activity were measured in GCF, before (day 0) and after treatment (7th and 30th day).

Antagonistically positioned healthy teeth were used as a control.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the condition of teeth:

* Presence of proximal caries on anterior and posterior teeth
* Existence of the antagonistic tooth ("mirror"-positioned healthy tooth) to be used as control
* An absence of fresh post-extraction or traumatic wounds in the restoration area or in the area of restored surfaces
* An absence of infection in the area of restored surfaces

Other influencing criteria:

* Absence of bone-associated diseases or treatments
* Satisfactory oral hygiene
* Patients exhibiting good compliance

Exclusion Criteria:

Criteria related to the condition of teeth:

* Endodontic and/or periodontal infections in the area of the cervical filling
* Presence of periodontopathy
* Prominent periodontal pockets
* Subgingival carries
* Prominent fillings outside the cavity

Other influencing criteria:

* Patients on radiation or immunosuppressive therapy
* Presence of bone-associated diseases and malignant diseases
* Patients using drugs/alcohol/cigarettes (> 20 cigarettes per day)
* Bad oral hygiene
* Patients exhibiting poor compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Changes in the levels of MDA in dental patients GCF after the applied treatments | 0th, 7th and 30th days.
  The concentration of MDA in GCF was measured before (0 day) and twice after the applied treatments (7th and 30th days). GCF was taken via the intracervical absorption technique. Control GCF (from mirror-positioned health teeth) was taken once before the treatment.

SECONDARY OUTCOMES:
Changes in the levels of GSH in dental patients GCF after the applied treatments | 0th, 7th and 30th days.
  Concentration of GSH in GCF was measured before (0 day) and twice after the applied treatments (7th and 30th days). GCF was taken via the intracervical absorption technique. Control GCF (from mirror-positioned health teeth) was taken once before the treatment.

OTHER OUTCOMES:
Changes in tSOD activity in dental patients GCF after the applied treatments | 0th, 7th and 30th days.
  Activity of tSOD was measured before (0 day) and twice after the applied treatments (7th and 30th days). GCF was taken via the intracervical absorption technique. Control GCF (from mirror-positioned health teeth) was taken once before the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjana M Djukic, PhD, Pharm., Principal Investigator — University of Belgrade; Danilo V Vojvodic, Study Director — Military Medical Academy, Belgrade
Locations (1):
- Military Medical Academy, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khurshid Z, Mali M, Naseem M, Najeeb S, Zafar MS. Human Gingival Crevicular Fluids (GCF) Proteomics: An Overview. Dent J (Basel). 2017 Feb 22;5(1):12. doi: 10.3390/dj5010012. PMID 29563418
- [Background] Stefanovic V, Taso E, Petkovic-Curcin A, Dukic M, Gardasevic M, Rakic M, Xavier S, Jovic M, Miller K, Stanojevic I, Vojvodic D. Influence of dental filling material type on the concentration of interleukin 9 in the samples of gingival crevicular fluid. Vojnosanit Pregl. 2016 Aug;73(8):728-34. doi: 10.2298/VSP140227054S. PMID 29328596
- [Background] Gaut JP, Byun J, Tran HD, Lauber WM, Carroll JA, Hotchkiss RS, Belaaouaj A, Heinecke JW. Myeloperoxidase produces nitrating oxidants in vivo. J Clin Invest. 2002 May;109(10):1311-9. doi: 10.1172/JCI15021. PMID 12021246
- [Background] Djukic MM, Jovanovic MD, Ninkovic M, Stevanovic I, Ilic K, Curcic M, Vekic J. Protective role of glutathione reductase in paraquat induced neurotoxicity. Chem Biol Interact. 2012 Aug 30;199(2):74-86. doi: 10.1016/j.cbi.2012.05.008. Epub 2012 Jun 18. PMID 22721943
- [Background] Begic A, Djuric A, Ninkovic M, Stevanovic I, Djurdjevic D, Pavlovic M, Jelic K, Pantelic A, Zebic G, Dejanovic B, Stanojevic I, Vojvodic D, Milosavljevic P, Djukic M, Saso L. Disulfiram moderately restores impaired hepatic redox status of rats subchronically exposed to cadmium. J Enzyme Inhib Med Chem. 2017 Dec;32(1):478-489. doi: 10.1080/14756366.2016.1261132. PMID 28102089
- [Background] Djuric A, Begic A, Gobeljic B, Pantelic A, Zebic G, Stevanovic I, Djurdjevic D, Ninkovic M, Prokic V, Stanojevic I, Vojvodic D, Djukic M. Subacute alcohol and/or disulfiram intake affects bioelements and redox status in rat testes. Food Chem Toxicol. 2017 Jul;105:44-51. doi: 10.1016/j.fct.2017.03.041. Epub 2017 Mar 24. PMID 28344087
- [Background] Nazar Majeed Z, Philip K, Alabsi AM, Pushparajan S, Swaminathan D. Identification of Gingival Crevicular Fluid Sampling, Analytical Methods, and Oral Biomarkers for the Diagnosis and Monitoring of Periodontal Diseases: A Systematic Review. Dis Markers. 2016;2016:1804727. doi: 10.1155/2016/1804727. Epub 2016 Dec 15. PMID 28074077